CLINICAL TRIAL: NCT06750939
Title: The Impact of Propofol and Ketamine on Cardiovascular Collapse During Induction for Endotracheal Intubation in Critically Ill Patients: A Prospective Observational Study
Brief Title: The Impact of Propofol and Ketamine on Cardiovascular Collapse During Induction for Intubation
Status: Recruiting | Type: Observational
Sponsor: Kocaeli City Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: ksh.Oemgin.001
Record Dates: First submitted 2024-12-05; First posted 2024-12-27 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Cardiovascular Collapse; Intubation Complication; Anaesthetic Complication Cardiac
Keywords: cardiac arrest; intubation; shock index
MeSH Terms: conditions — Shock; Heart Arrest | interventions — Propofol; Ketamine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cardiovascular collapse: "- At least one documented episode of SpO₂ < 80%, ensuring accuracy of measurement.
  * At least one episode of systolic arterial blood pressure (SAB) < 65 mmHg.
  * SAB < 90 mmHg sustained for a duration of 30 minutes.
  * Initiation of norepinephrine therapy.
  * Escalation of pre-existing norepinephrine infusion dose.
  * Administration of >15 mL/kg crystalloid fluids to achieve SAB > 90 mmHg.
  * Occurrence of cardiac arrest." The occurrence of any of the above-mentioned events within the first 30 minutes following the initiation of the intervention will be considered as cardiovascular collapse.
  Interventions: Other: propofol; Other: ketamine
- No Cardiovascular collapse
  Interventions: Other: propofol; Other: ketamine

INTERVENTIONS:
Other: propofol — The hemodynamic effects of propofol and ketamine are well-documented in the general patient population, yet the incidence and characteristics of cardiovascular collapse induced by these agents in critically ill patients remain underexplored. Cardiovascular collapse, a severe and potentially life-threatening event, may arise due to the unique physiological stressors present in the critical care setting, including pre-existing hemodynamic instability, comorbidities, and the administration of high-risk pharmacological agents. Despite the theoretical understanding of these drugs' pharmacodynamics, there is limited evidence assessing their differential impact on cardiovascular function in this vulnerable population.
  This study aims to contribute novel insights to the literature by exploring the association between these widely used sedative-hypnotic agents and the development of cardiovascular collapse. While propofol is known for its potent vasodilatory and myocardial depressive effects,
Other: ketamine — The hemodynamic effects of propofol and ketamine are well-documented in the general patient population, yet the incidence and characteristics of cardiovascular collapse induced by these agents in critically ill patients remain underexplored. Cardiovascular collapse, a severe and potentially life-threatening event, may arise due to the unique physiological stressors present in the critical care setting, including pre-existing hemodynamic instability, comorbidities, and the administration of high-risk pharmacological agents. Despite the theoretical understanding of these drugs' pharmacodynamics, there is limited evidence assessing their differential impact on cardiovascular function in this vulnerable population.
  This study aims to contribute novel insights to the literature by exploring the association between these widely used sedative-hypnotic agents and the development of cardiovascular collapse. While propofol is known for its potent vasodilatory and myocardial depressive effects,

SUMMARY:
This prospective observational study evaluates the impact of propofol and ketamine on the risk of cardiovascular collapse during induction for endotracheal intubation in critically ill patients. Induction agents play a crucial role in managing hemodynamic stability, particularly in this vulnerable population. Propofol, known for its vasodilatory and myocardial depressant effects, has been associated with significant hypotension during induction. Conversely, ketamine, with its sympathomimetic properties, is often considered a safer alternative for hemodynamic stability.

In addition to comparing the incidence of cardiovascular collapse-defined as severe hypotension or cardiac arrest-this study examines the relationship between these induction agents and shock indices, including systolic shock index, diastolic shock index, age-adjusted shock index, and modified shock index. These parameters will provide a more detailed understanding of the hemodynamic effects of each agent and their clinical implications. The findings aim to guide induction agent selection to optimize outcomes in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Patients admitted to the intensive care unit (ICU) who undergo endotracheal intubation during their ICU stay will be included.

Exclusion Criteria:

* Patients who did not provide consent to participate in the study
* Patients intubated due to cardiac arrest
* Patients intubated outside the intensive care unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit (ICU) who undergo endotracheal intubation during their ICU stay will be included.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
cardiovascular collapse | The occurrence of any of the above-mentioned events within the first 30 minutes following the initiation of the intervention will be considered as cardiovascular collapse.
  * At least one documented episode of SpO₂ < 80%, ensuring accuracy of measurement.
  * At least one episode of systolic arterial blood pressure (SAB) < 65 mmHg.
  * SAB < 90 mmHg sustained for a duration of 30 minutes.
  * Initiation of norepinephrine therapy.
  * Escalation of pre-existing norepinephrine infusion dose.
  * Administration of >15 mL/kg crystalloid fluids to achieve SAB > 90 mmHg.
  * Occurrence of cardiac arrest.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli City Hospital, Köseköy, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We regret to inform that the data from this study will not be shared due to constraints related to authorization and time limitations. However, those interested may contact the study's corresponding author to request access to the data.